CLINICAL TRIAL: NCT01663064
Title: Zenith® p-Branch™: Single-Center Study
Acronym: PBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-018
Record Dates: First submitted 2012-08-02; First posted 2012-08-13 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Aortic Aneurysm; Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm; Endovascular; Fenestration; Juxtarenal; Off-the-shelf; Pararenal
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Abdominal

ARMS (1):
- Endovascular (Experimental): Endovascular treatment
  Interventions: Device: Endovascular treatment (Zenith® p-Branch™ endovascular graft)

INTERVENTIONS:
Device: Endovascular treatment (Zenith® p-Branch™ endovascular graft) — Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guides the study device(s) into place in the aorta.

SUMMARY:
The Zenith® p-Branch™: Single-Center Study is a clinical trial approved by Swedish Regulatory Authority to study the safety and effectiveness of the Zenith® p-Branch™ in the treatment of abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Pararenal or juxtarenal AAA >5.0 cm in diameter
* Pararenal or juxtarenal AAA with history of growth >0.5 cm/year

Exclusion Criteria:

* Age < 18 years
* Life expectancy < 2 years
* Pregnant or breast feeding
* Inability or refusal to give informed consent by the patient or a legally authorized representative
* Unwilling or unable to comply with the follow-up schedule
* Additional medical restrictions as specified in the Clinical Investigation Plan
* Additional anatomical restrictions as specified in the Clinical Investigation Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-06; Primary Completion 2015-10 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Technical Success | Up to 5 years
  Technical success is described as: 1) successful access of the aneurysm site, 2) successful deployment of the Zenith® p-Branch™ endovascular graft in the intended location, 3) Zenith® p-Branch-™ endovascular graft is patent at deployment completion as evidenced by intraoperative angiography, and 4) all vessels targeted with a fenestration are patent at deployment completion as evidenced by intraoperative angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A. Resch, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skane University Hospital, Malmo, Sweden